CLINICAL TRIAL: NCT04028232
Title: Influence of Socio-Economic Factor on Net Survival in Patients With Multiple Sclerosis in France ( ECOVIMUS).
Acronym: ECOVIMUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Ecole des Hautes Etudes en Santé Publique (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 18512
Record Dates: First submitted 2019-07-19; First posted 2019-07-22 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: C10.114.375.500
Keywords: Multiple Sclerosis; Epidemiology; Socio-Economic Status; Net Survival
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: In comparison to general population, persons with Multiple Sclerosis have a higher risk to premature death with an estimate reduced life expectancy from 7 to 14 years. However, risk factors of mortality in MS are not well identified and well known. Following the example of studies carry on cancers survival, socioeconomic status (SES) may have an influence on survival in MS.

Objective: The main objective of ECOVIMUS is to estimate net survival according to SES using the European Deprivation Index as a proxy and other major covariates (gender, initial clinical phase and years of disease onset).

Methods: In order to answer to our main objective, we will use a retrospective cohort of MS patients with a medical follow-up in one of the 18 centers included in SURVIMUS II, with a MS onset between 1960 and 2015 and with an informed vital at the date of December 31st, 2015.

The ecological score of deprivation EDI will be used as a proxy of the socioeconomic status and will be attributed from the geolocalisation to patient's residence address. Net survival is directly associated to the notion of "mortality in excess". This mortality will be estimated comparing the observed mortality in MS patients to mortality in the general population. The advantage of this methodological approach is that cause of death is not needed.

Statistical analysis: The influence of socioeconomic status on the excess of mortality will be estimated thanks to a parametric multivariate model of excess rate mortality. This model will be adjusted on other major covariates (gender, age at disease onset, and initial clinical phase) and will include potential complex effects as non-linearity, non-proportionality and interactions.

Expected results: We expect to highlight some differences of net survival in MS patients according to socioeconomic group as it was already shown in cancers. This study will complete information on factors of mortality excess in MS and knowledge on socioeconomic inequalities encountered all along MS disease course.

ELIGIBILITY:
Inclusion Criteria:

* all patients registered in 17 selected French OFSEP centres with core dataset with a sufficient level of data
* Diagnosis a of definite or probably MS according to Poser or McDonald criteria. With an MS onset date between January 1st, 1960 and December 31st, 2015.
* With a postal residence address well informed in the OFSEP database.

Exclusion Criteria:

* MS patients with less than one year's disease duration by the study end will be excluded.

Ages: 1 Year to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include all patients registered in 17 selected French OFSEP centres with core dataset with a sufficient level of data (Besançon, Bordeaux, Caen, Clermont-Ferrand, Dijon, Lille, Lyon, Marseille, Nancy, Nice, Rennes, Saint-Etienne, Strasbourg, Toulouse, Montpellier, Nantes, Nîmes). The minimum required data includes: Diagnosis a of definite or probably MS according to Poser or McDonald criteria. With an MS onset date between January 1st, 1960 and December 31st, 2015. With a postal residence address well informed in the OFSEP database.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Excess mortality survival | From date of MS onset to the date of patients death or to study cut-off date on 1st January 2016.
  Net survival is defined as the probability of death in a hypothetical setting where the cause of interest (in our case MS) would be the only possible cause of death. It is directly linked to the concept of the "excess mortality due to the studied disease". Net survival can be calculated according to two settings, either the estimator of survival can be calculated from death due to MS while cause of death are known, either it can be calculated from the excess of mortality due to MS compared to the mortality of the general population obtained from mortality table of the generable population.

SECONDARY OUTCOMES:
European Deprivation Index (EDI) proxy of Socio-Economic Status | From date of MS onset to the date of patients death or to study cut-off date on 1st January 2016.
  The EDI Score is a combination of weighted ecological variates and is available for each 'IRIS area' (Ilots regroupés pour l'Information Statistique). An IRIS area represents the smallest geographical entity for which census data are available in France.
  The geolocation of each individual address, according to latitude and longitude coordinates, is performed with the system of geographical information (SGI) ARGIS® 10.5. This point of geolocation is correlated to the IRIS area and then an EDI score can be attributed to patients registered in the database. The EDI score can be categorized into quintiles.
Distance to MS expert care center | From date of MS onset to the date of patients death or to study cut-off date on 1st January 2016.
  Distance in kilometer by road transport from residence place to MS expert care center

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - University Hospital Center of CAEN, Caen, Normandy
  - University Hospital of Besancon, Besançon
  - University Hospital of Bordeaux, Bordeaux
  - University Hospital Centre of Caen, Caen
  - University Hospital of Clermont Ferrand, Clermont-Ferrand
  - University Hospital of Dijon, Dijon
  - University Hospital of Lille, Lille
  - University Hospital of Lyon, Lyon
  - University Hospital of Marseille, Marseille
  - University Hospital of Montpellier, Montpellier
  - University Hospital of Nancy, Nancy
  - University Hospital of Nantes, Nantes
  - University Hospital of Nice, Nice
  - University hospital Centre of Nîmes, Nîmes
  - University Hospital of Rennes, Rennes
  - University Hospital Centre of Saint-Etienne, Saint-Etienne
  - University Hospital of Strasbourg, Strasbourg
  - University Hospital Centre of Toulouse, Toulouse